CLINICAL TRIAL: NCT03132090
Title: Early Response Monitoring of Systemic Therapies in Patients With Advanced Melanoma by Simultaneous Positron-emission-tomography (PET)/Magnetic Resonance Imaging (MRI)
Brief Title: Early Therapy Response Monitoring in Melanoma Patients Using PET/MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Nina Schwenzer, Prof. Dr. med. Nina Schwenzer (clinical professor & PI), University Hospital Tuebingen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GK-MR/PET Tü-004
Record Dates: First submitted 2017-03-07; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Malignant Melanoma Stage IV
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/MR (Biograph mMR) — The combination of PET and MRI allows for evaluation of metabolic, functional and morphological parameters such as glucose metabolism, perfusion, diffusion restriction or size in one examination. Due to the combination of MRI and PET in one scanner it is possible to align the acquired PET and MR datasets with high precision

SUMMARY:
Therapeutic agents used in malignant melanoma treatment such as BRAF/MEK inhibitors and anti-CTLA-4/Anti-PD-1 antibodies go along with harmful side effects in a considerable proportion of patients and treatment costs may cause relevant medical expenditures per month. Currently, therapy response assessment in melanoma patients is performed using RECIST criteria which are based on changes in tumour size. PET/CT combines morphological and metabolic information. Thus, the so-called PERCIST-criteria were introduced integrating change in size and glucose utilization for response assessment in solid tumors. Due to the different mechanism of action these new agents introduce different response patterns increase in tumor size due to inflammation for antibody therapies). In conventional chemotherapies, re-staging is usually performed 3 months after treatment initiation which is the result of empirical investigations. Moreover, it has recently been shown, that response to new targeted therapies can be detected much earlier using PET or functional MR techniques. This forms the rationale for the monitoring of melanoma patients using a combined PET/MR technique after only 2 weeks of therapy initiation. Especially for patients in stage IV with a medium survival time of 12 months, a 2.5 months earlier re-staging and therapy adjustment would have significant consequences for the individual clinical course.

ELIGIBILITY:
Inclusion Criteria:

* patient with diagnosed unresectable malignant melanoma stage IV
* age: ≥18 years
* planned systemic therapy with either new therapies (BRAF/MEK inhibitors, Anti-CTLA-4/Anti-PD-1 antibodies) or conventional chemotherapeutics (CTx)
* clinically indicated routine PET/CT (baseline t0) demonstrating at least one measurable lesion
* PET/CT for baseline-staging and therapy monitoring (clinical indication required)
* informed consent

Exclusion Criteria:

* contraindications for MR-imaging (metal implants, claustrophobia, etc.)
* contraindications for gadolinium-based contrast agent
* acute infections or other acute diseases
* pregnant or breast-feeding women
* disability for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2014-09-29 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Early therapy response assessment | Baseline t0 (1st imaging / start of therapy), early therapy response (study visit) t1 (2 weeks after therapy start), regular therapy response (routine visit) t2 (3 month after therapy start)
  Early therapy response assessment by multiparametric hybrid imaging (PET/MRI) two weeks (early time point - study visit) and three months (regular staging) after therapy initiation with regard to optimizing patient management (please note: no therapy change intended based on the imaging at early time point (study visit t1)). Early study imaging data and later regular imaging data have to be compared.

SECONDARY OUTCOMES:
prognostic capacity of morphological and functional MRI measures | 3 month
  testing the prognostic capacity of morphological and functional MRI measures (diffusion, perfusion) for predicting the concordance of therapy response results two weeks and three months after treatment initiation
prognostic value of PET/MRI-specific response | 18 month
  validation of the significance and prognostic value of the defined PET/MRI-specific response evaluation criteria by correlation with TTP

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Radiology, University of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seith F, Forschner A, Weide B, Guckel B, Schwartz M, Schwenck J, Othman AE, Fenchel M, Garbe C, Nikolaou K, Schwenzer N, la Fougere C, Pfannenberg C. Is there a link between very early changes of primary and secondary lymphoid organs in 18F-FDG-PET/MRI and treatment response to checkpoint inhibitor therapy? J Immunother Cancer. 2020 Aug;8(2):e000656. doi: 10.1136/jitc-2020-000656. PMID 32753543